CLINICAL TRIAL: NCT04717570
Title: Early Feasibility Study for the Foldax TRIA Mitral Heart Valve Replacement Investigational Device Exemption
Brief Title: Early Feasibility Study for the Foldax TRIA Mitral Heart Valve Replacement
Acronym: FOLDAX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foldax, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Foldax CP-002
Record Dates: First submitted 2020-12-14; First posted 2021-01-22 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Mitral Valve Disease; Mitral Valve Stenosis; Mitral Valve Failure
MeSH Terms: conditions — Mitral Valve Stenosis

STUDY DESIGN:
Intervention Model Description: All patients will receive the study device
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- TRIA Mitral Valve (Experimental): Patients receiving the Foldax Mitral Valve
  Interventions: Device: Foldax TRIA Mitral Valve

INTERVENTIONS:
Device: Foldax TRIA Mitral Valve — Mitral Valve Replacement

SUMMARY:
The purpose of this study is to conduct the initial clinical investigation of the Foldax Polymer Mitral Valve to collect evidence on the device's safety and performance. The study is anticipated to confirm successful clinical safety and clinical effectiveness with significant improvements in clinical hemodynamic performance.

DETAILED DESCRIPTION:
The Foldax Polymer Mitral Valve is indicated as a replacement for a diseased, damaged, or malfunctioning native mitral heart valve via open heart surgery. This is a first in human study conducted under US FDA's Early Feasibility Investigational Device Exemption and will enroll up to 15 patients. These patients will be followed up to 5 years after implantation.

ELIGIBILITY:
Inclusion Criteria:

* Is 18 years or older
* Is a candidate for mitral valve replacement with cardiopulmonary bypass
* Is a candidate for mitral valve replacement due to:
* Moderate to severe mitral valve stenosis,
* Moderate to severe mitral valve regurgitation, or
* Moderate to severe mixed mitral stenosis/regurgitation
* Able to withstand short term anticoagulation
* Willing and able to comply with protocol requirements

Exclusion Criteria:

* Prior mitral valve surgery for valve replacement or valve repair (this does NOT include percutaneous interventions i.e. Mitraclip, chordal replacement)
* Requires emergency surgery
* Requires other planned surgery within 12 months of valve replacement
* Active endocarditis or active myocarditis
* Acute preoperative neurological deficit defined as neurological deficit < 3 months prior to enrollment
* Non-cardiac illness resulting in a life expectancy of less than 12 months
* Enrolled in another investigational device or drug study (enrolled patients may not enroll in other studies)
* Myocardial infarction, or severe cardiac adverse event which has not returned to baseline for at least 30-days prior to enrollment
* Aortic aneurysm or other medical condition that creates a higher than usual risk of surgical complications
* Renal or hepatic failure
* Hematological disorders, patients must not have a hematocrit of <30%, hemoglobin <10 g/dL, platelet count of <100,000 cells/µL, or WBC <4,000 cells/µL; coagulation profile must not be outside of normal limits
* Patients who are prisoners or mentally ill
* Patients who are pregnant or expect to become pregnant in the 12 months following implantation, or are lactating
* Has a positive test result for COVID-19 virus (baseline or preoperative)
* Patients who have withdrawn after implantation may not re-enter
* Intraoperatively it is determined that the patient anatomy is not compatible with the device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoints | 12 months following patient enrollment completion
  Adverse Event (AE) rates for valve related early and late complications : thromboembolism, valve thrombosis, major hemorrhage, major paravalvular leak, endocarditis, structural valve deterioration, nonstructural valve dysfunction, valve related hemolysis, all cause death, valve related reoperation, valve explant, and valve related death. Results are visually compared to event rates reported in the literature.
Primary Effectiveness Endpoints- Change in Hemodynamic Performance | 12 months following patient enrollment completion
  Hemodynamic performance parameters are mmHG mean gradient and derived Effective Orifice Area (EOA). Success is defined as clinically significant improvement in hemodynamic performance (Effective Orifice Area (EOA)) at one year based on literature reports for surgical aortic valve replacement.
Clinical Effectiveness: Change in New York Heart Association Assessment | 12 months following patient enrollment completion
  Clinically significant improvement (one grade) in the New York Heart Association (NYHA) functional classification status at 365 days compared to baseline. a. Class I - No symptoms and no limitations in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc. b. Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity. c. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100m). Comfortable only at rest. d. Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.

SECONDARY OUTCOMES:
Number of Participants with Stroke | 5 years following patient enrollment
  Assessment of patient experiencing a stroke (ex; ischemic stroke, intracerebral hemorrhage, subarachnoid hemorrhage, or other) verified by imaging and or physical exam
Number of Participants with Transient Ischemic Attack | 5 years following patient enrollment
  Assessment of patient having a TIA as verified by imaging and or physical exam
Number of Participants with Migration of the TRIA valve | 5 years following patient enrollment
  Assessment of patient experiencing valve migration as verified by imaging, procedure, or physical exam.
ICU Duration of Stay | 30 days post patient enrollment
  Length of stay in the ICU post valve implantation defined as arrival time/date in hours and minutes to transfer to floor time/date in hours and minutes.
Ventilation Time | 30 days post patient enrollment
  Ventilation time in hours defined as arrival time/date in recovery in hours and minutes to date and time extubated in hours and minutes
New Onset Atrial Fibrillation | 12 months post patient enrollment
  New/post-operative atrial fibrillation - confirmed on ECG after closure during initial or subsequent admission or at one-year review
Readmission within 30 days of discharge | 30 days post patient discharge date
  Patient readmission to the hospital post discharge measured by date/time
Post Procedure length of stay | 30 days post patient enrollment
  l. Post procedure length of stay defined as the time/date documented for arrival in the recovery unit to date/ time of discharge in hours and minutes.
Kansas City Cardiomyopathy Questionnaire (KCCQ) | 12 months post patient enrollment
  Change in QOL as measured by the KCCQ. Scores are measured from 0-100, in hich higher scores reflect better health status.
Six Minute Walk Test | 12 months post patient enrollment
  Change in patients activity tolerance as documented by a 6 Minute Walk Test assessed by distance traveled after 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Frank Shannon, MD, Study Chair — Beaumont Hospital
Locations (3):
- United States (3):
  - St. Vincent Hospital, Carmel, Indiana
  - Ascension Via Christi St. Francis, Wichita, Kansas
  - The Christ Hospital, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No